CLINICAL TRIAL: NCT00791817
Title: An Open-label, Single Dose, Randomized, Crossover Study to Evaluate Potential Food Effects
Brief Title: Study to Evaluate Potential Food Effects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: William S Aronstein, PhD, MD, Procter and Gamble Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2005046B
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Results first posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: pharmacokinetics study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 200 mg PG 760564, Subjects Fasted (Experimental): 200 mg PG 760564, Subjects Fasted, single dose
  Interventions: Drug: PG-760564
- 200 mg PG 760564, Subjects Fed (Experimental): 200 mg PG 760564, Subjects Fed high fat meal
  Interventions: Drug: PG-760564

INTERVENTIONS:
Drug: PG-760564 — 200 mg capsule, single dose,fasted when dosed, duration is 4 days
  Arms: 200 mg PG 760564, Subjects Fasted
Drug: PG-760564 — 200 mg capsule, single dose,high fat diet when dosed, duration is 4 days
  Arms: 200 mg PG 760564, Subjects Fed

SUMMARY:
Half the group will be given a high fat diet and the other half will fast. They will then be crossed over.

DETAILED DESCRIPTION:
A food-effect study which will be conducted at any time during the MRD study period on one single cohort of subjects using 200 mg oral dose of PG 760564. Half the group will be given a high fat diet and the other half will fast. They will ten be crossed over.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and surgically sterile or post-menopausal (last menstrual period > 1 year at the time of enrollment) healthy females, 18-45 years of age, inclusive, at screening;
* Who have not used tobacco or nicotine-containing products within the past 3 months;
* Willing to abstain from caffeine or xanthine-containing beverages, including coffee and tea, chocolate, alcohol, grapefruit juice, and Seville oranges, from 24 hours before admission and for the duration of the study;
* Who have a body mass index (BMI) between 18 and 32 kg/m2, inclusive.

Exclusion Criteria:

* History of diabetes, cardiovascular, hepatic, renal, or malabsorptive disease;
* History of diabetes, cardiovascular, hepatic, renal, or malabsorptive disease;
* History of peptic ulcer disease, hemorrhoids, GI surgery (appendectomy and cholecystectomy are allowed), or GI bleeding;
* History of autoimmune disease;
* History of immunodeficiency or of unusual susceptibility to infectious diseases;
* History of tuberculosis, acquired immunodeficiency syndrome (AIDS), or infection with human immunodeficiency virus (HIV);
* Any history of hypersensitivity or clinically significant allergy to any drug;
* Personal or family history of prolonged QT syndrome or any cardiac conduction abnormality;
* Family history of sudden death;
* History of uveitis or inflammatory ocular disease;
* History of peptic ulcer disease, hemorrhoids, GI surgery (appendectomy and cholecystectomy are allowed), or GI bleeding;
* History of autoimmune disease;
* History of immunodeficiency or of unusual susceptibility to infectious diseases;
* History of tuberculosis, acquired immunodeficiency syndrome (AIDS), or infection with human immunodeficiency virus (HIV);
* Any history of hypersensitivity or clinically significant allergy to any drug;
* Personal or family history of prolonged QT syndrome or any cardiac conduction abnormality;
* Family history of sudden death;
* History of uveitis or inflammatory ocular disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2005-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William S Aronstein, MD, PhD, Study Director — Procter and Gamble
Locations (1):
- Stuart I Harris, MD, PhD, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 200 mg PG 760564. Fed Then Fasted: 200 mg PG 760564. subjects dosed in a Fed State, followed by a washout period, followed by 200 mg PG 760564 in a fasted state
- 200 mg PG 760564. Fasted: 200 mg PG 760564. subjects dosed in a Fasted , followed by a washout period, followed by 200 mg PG 760564 in a Fed state
Period: 1: Single Dose Followed by Week Washout
Arm/Group | 200 mg PG 760564. Fed Then Fasted | 200 mg PG 760564. Fasted
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: 2: Single Dose
Arm/Group | 200 mg PG 760564. Fed Then Fasted | 200 mg PG 760564. Fasted
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 mg PG 760564. Fed Then Fasted | 200 mg PG 760564. Fasted | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] — Study is a crossover study. All subjects received Investigational Product in BOTH the Fed and Fasted state
  years | 31.8 (10.0) | 31.8 (10.0) | 31.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum plasma concentration after a single dose
Time Frame: over 12 hours
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | 200 mg PG 760564. Fed Then Fasted | 200 mg PG 760564. Fasted
Number analyzed (Participants) | 10 | 10
ng/mL | 2567.9 (652.6) [1.20 to 1.61] | 3568.9 (633.2) [1.20 to 1.61]
Statistical Analysis 1: Comparison: 200 mg PG 760564. Fed Then Fasted vs 200 mg PG 760564. Fasted; values are Geometric Means and Confidence Intervals are on the Ratio of Fed to Fasted; Test type: Superiority or Other; Confidence Interval is on the Ratio of Fed to Fasted; Mean Difference (Net) = 1.3897, 90% CI 2-sided [1.1998 to 1.6097] — Confidence Interval is on the Ratio of Fed to Fasted

ADVERSE EVENTS:
Arm/Group | 200 mg PG 760564. Fed Then Fasted | 200 mg PG 760564. Fasted
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg PG 760564. Fed Then Fasted (N=10) | 200 mg PG 760564. Fasted (N=10)
heme-positive stool (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data, calculations, interpretations, opinions, and recommendations are the property of P&GP. In the event study results are published in the scientific literature by P&GP, acknowledgment will be made to the Investigator(s) in the accepted style, as appropriate.